CLINICAL TRIAL: NCT06371053
Title: The Effect of Community Intervention on Different Degrees of Dementia: A Randomized Controlled Study
Brief Title: The Effect of Community Intervention on Different Degrees of Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babujinaya Cela (Other Government)
Responsible Party: Sponsor-Investigator, Babujinaya Cela, Research Director, Buraidah Central Hospital
Organization: Buraidah Central Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: community - dementia
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): The elderly individuals will be arranged to undergo a continuous three-week (21 days) duration of Community Intervention, with weekends off and training conducted only on weekdays, two sessions per day, each lasting 15-20 minutes.
  Interventions: Behavioral: Community Intervention
- the blank group (No Intervention): No intervention will be applied

INTERVENTIONS:
Behavioral: Community Intervention — The intervention includes Cognitive Training: Activities targeting memory, attention, language, and executive functions to maintain cognitive abilities. This could involve cognitive games, memory exercises, and daily tasks.
  Life Skills Training: Assistance in maintaining or relearning daily life skills such as personal hygiene, dressing, eating, and household chores. This could be through structured training programs and daily guidance.
  Physical Exercise: Providing appropriate physical activities and exercises to maintain physical health and function, including walking, balance training, and light strength training.
  Social Support: Organizing social activities and support groups to facilitate interaction and reduce social isolation and loneliness.
  Emotional Support: Offering mental health support and psychosocial services to help individuals cope with emotional challenges such as anxiety and depression.
  Arms: the intervention group

SUMMARY:
The goal of this clinical trial is to explore the impact of Community Intervention on Dementia and Activities of Daily Living in community-dwelling elderly individuals (≥60 year old) with Alzheimer's disease. It primarily aims to address: the effects of Community Intervention on Dementia and Activities of Daily Living in community-dwelling elderly individuals with Alzheimer's disease in different degrees. All participants are required to undergo a continuous 2-week (14 days) Community Intervention, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 30 minutes each.

DETAILED DESCRIPTION:
Regular exercise can increase brain function, improve memory, speed up cognitive processes, and fight off diseases like Alzheimer ' s and dementia.

The goal of this clinical trial is to explore the impact of Community Intervention on Dementia and Activities of Daily Living in community-dwelling elderly individuals (≥60 year old) with Alzheimer's disease. It primarily aims to address: the effects of Community Intervention on Dementia and Activities of Daily Living in community-dwelling elderly individuals with Alzheimer's disease in different degrees. All participants are required to undergo a continuous 2-week (14 days) Community Intervention, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 30 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years old.
* No hospitalization within the past six months.
* Alzheimer's disease
* The elderly people who voluntarily participate and agree to adhere until the end of the study.

Exclusion Criteria:

* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Physical disability.
* Difficulty in mobility.
* Simultaneously receiving other therapies that might influence this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | day 1 and day 14
  The Mini-Mental State Examination (MMSE) is a widely used tool for assessing cognitive function, particularly in the elderly population. It evaluates various cognitive domains such as orientation, memory, attention, calculation, and language.
  The test consists of a series of questions and tasks, including asking the individual to state the current date, recall a list of words, perform simple calculations, and follow verbal commands. Each correct response earns a certain number of points, and the total score ranges from 0 to 30, with higher scores indicating better cognitive function.

SECONDARY OUTCOMES:
Barthel Index | day 1 and day 14
  The Barthel Index is a scale used to measure a person's ability to perform activities of daily living. It was developed by Dr. Mahlon R. Barthel in the 1960s and has since been widely used in healthcare settings, particularly in rehabilitation and geriatric care. The scores range between 0 and 100, with higher scores indicating better activities of daily living.
Functional near-infrared spectroscopy | day 1 and day 14
  Functional near-infrared spectroscopy (fNIRS) is a non-invasive neuroimaging technique that measures changes in cerebral blood oxygenation and hemodynamics. It provides a way to monitor brain activity by measuring the concentration changes of oxygenated hemoglobin (HbO) and deoxygenated hemoglobin (HbR) in the cortical tissue. The numerical values displayed by near-infrared will be recorded, with higher values indicating more active brain blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Wi, Principal Investigator — Site Coordinator of United Medical Group

IPD SHARING:
Plan to Share IPD: No